CLINICAL TRIAL: NCT06323200
Title: The Impact of Surgical Intervention on Lymphatic System in Patients With Lymphedema
Brief Title: Lymphedema Duration on Lymphatic Vessel Quality and Outcomes After LVA
Acronym: LVA
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202400221B0
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Lymphedema
Keywords: retrospective cohort
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lymphedema duration > 3.6 years
  Interventions: Procedure: lymphaticovenous anastomosis
- Lymphedema duration ≤ 3.6 years
  Interventions: Procedure: lymphaticovenous anastomosis

INTERVENTIONS:
Procedure: lymphaticovenous anastomosis — The patients were under intravenous general anesthesia with local anesthetic infiltration for each incision21. LVs were detected by intradermal injection of ICG into the web spaces between the toes and on the medial and lateral malleoli. ICG flow with linear dermal backflow(DB) patterns was detected immediately using a handheld near-infrared camera. The recipient veins were marked using B-mode echo Doppler, close to the marked linear pattern. In case of DB pattern, the incision was made along the great saphenous vein. A 3 cm incision was made and the lymphatics and recipient veins were identified. All patients underwent supermicrosurgical LVA with 11- 0 nylon sutures using a high-power surgical microscope by a single senior surgeon. LVAs are performed using only antegrade flow lymphatics and lymphaticovenous end-to-end anastomosis (LVEEA) and end-to-side anastomosis (LVESA).

SUMMARY:
This study aimed to address the impact of lymphedema duration on the quality of lymphatic vessels as well as the outcome after LVA using propensity score matching.

DETAILED DESCRIPTION:
With an increase in the incidence and treatment of breast and gynecological cancers, an increase in the prevalence of secondary lymphedema has been witnessed1. As a consequence of lymphadenectomy and adjuvant radiotherapy, swollen limbs result from the accumulation of protein rich fluid2. Lymphedema is predicted to arise in 20-40% of patients with cervical and breast cancer3, which is a chronic disease that can significantly hamper quality of life4-6. Affected limbs may suffer from lifelong swelling with functional impairment and repeated cellulitis, and some may eventually progress to late-stage diseases such as elephantiasis and lymphorrhea7-9.

Supermicrosurgical lymphaticovenous anastomosis (LVA) is a well-documented minimally invasive treatment modality that bypasses lymph into the venous system to alleviate lymphedema10-14. It was a common belief that a longer lymphedema duration (LD) may be associated with inferior lymphatic vessel (LVs) quality, as well as excess fibrous components in the affected limbs, which are characteristics of advanced lymphedema. Consequently, owing to inferior LV quality, LVA is considered unsuitable for advanced cases; instead, vascularized lymph node transfer (VLNT) or excisional procedures are recommended7,15.

However, growing evidence has demonstrated the effectiveness of LVA for the treatment of severe lymphedema16-19. These findings, contrary to common beliefs, raise questions regarding the association between LD, LV quality, and outcomes after LVA. This study aimed to address the impact of LD on the quality of LV as well as the outcome after LVA using propensity score matching.

ELIGIBILITY:
Inclusion Criteria:

* This study including patients diagnosed with lymphatic-related diseases at Kaohsiung Chang Gung Memorial Hospital from September 2015 to March 2023.

Patients who underwent LVA for unilateral lower-limb lymphedema.

Exclusion Criteria:

* Primary lymphedema, bilateral lower limb lymphedema, history of previous LVA, vascularized lymph node transfer (VLNT), liposuction, or excisional therapy such as the Charles procedure, and those that were lost to follow-up.

Ages: 20 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients (age >20 years) receiving LVA for lower limb lymphedema at a tertiary medical center were retrospectively reviewed from September 2015 to March 2023.
Sampling Method: Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2023-03 (Actual); Study Completion 2023-03 (Actual)

PRIMARY OUTCOMES:
Volume change after LVA. | 6/12 months
  The primary endpoint was the volume change at 6/12 months after LVA.